CLINICAL TRIAL: NCT04445844
Title: IRENE Study: Phase 2 Study of INCMGA00012 and the Oncolytic Virus Pelareorep in Metastatic Triple Negative Breast Cancer
Brief Title: INCMGA00012 and Pelareorep for the Treatment of Metastatic Triple Negative Breast Cancer, IRENE Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mridula George, MD (Other)
Collaborators: Incyte Corporation (Industry); Oncolytics Biotech (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mridula George, MD, Assistant Professor of Medicine - Medical Oncology, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042001; NCI-2020-02940 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2020000268; Pro2020000268 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Breast Carcinoma; Metastatic Triple-Negative Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8; Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pelareorep, retifanlimab) (Experimental): Patients receive pelareorep IV over 60 minutes on days 1, 2, 15, and 16. Patients also receive INCMGA00012 IV over 60 minutes on day 3. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pelareorep; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Retifanlimab

INTERVENTIONS:
Biological: Pelareorep — Given IV
  Other Names: PO BB0209; PO-BB0209; Reolysin; Reovirus Serotype 3; Wild-type Reovirus
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Retifanlimab — Given IV
  Other Names: INCMGA 0012; INCMGA-0012; INCMGA00012; INCMGA0012; MGA 012; MGA-012; MGA012

SUMMARY:
This is a phase 2 study to evaluate the safety and efficacy of the combination of INCMGA00012 and pelareorep and to see how well they work in treating patients with triple negative breast cancer that has spread to other parts of the body (metastatic).

INCMGA00012 is a monoclonal antibody that works by attaching to the programmed cell death protein 1 (PD-1) and blocking this pathway, allowing the immune system to recognize and attack the cancer cells. Pelareorep is a type of virus called reovirus which occurs naturally and may break down cancer cells. Giving INCMGA00012 and pelareorep may slow the growth and spread of the cancer to another part of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of the combination of retifanlimab (INCMGA00012) and pelareorep for patients with metastatic triple negative breast cancer in the second and third line setting.

II. To assess the safety, tolerability and feasibility of INCMGA00012 in combination with the oncolytic virus pelareorep for patients with metastatic triple negative breast cancer in the second and third line setting.

SECONDARY OBJECTIVES:

I. To assess progression free survival (PFS), overall survival (OS) and duration of response (DOR) in patients receiving INCMGA00012 in combination with the oncolytic virus pelareorep for patients with metastatic triple negative breast cancer in the second and third line setting.

II. To assess quality of life measures.

EXPLORATORY OBJECTIVES:

I. To assess whether pre-treatment PD-L1 expression is associated with treatment outcomes.

II. To determine if changes in T cell repertoire as measured by T-cell receptor (TCR) sequencing is predictive of treatment outcomes.

OUTLINE:

Patients receive pelareorep intravenously (IV) over 60 minutes on days 1, 2, 15, and 16. Patients also receive retifanlimab IV over 60 minutes on day 3. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or inoperable locally advanced, histologically documented triple negative breast cancer (TNBC) (negative expression of estrogen receptor [ER], progesterone receptor [PR] and human epidermal growth factor receptor 2 [HER2] immunohistochemistry [IHC] 0 or 1+, HER2 fluorescence in situ hybridization [FISH] negative if IHC 2+, per American Society of Clinical Oncology [ASCO] College of American Pathologists [CAP] guidelines)
* Pre-menopausal and post-menopausal women who have received 1-2 prior lines of systemic therapy for metastatic triple negative breast cancer. Patients must have received at least one prior line of chemotherapy
* Patients who have received adjuvant therapy for locally advanced triple negative breast cancer may be eligible for the study if they relapse with metastatic disease within 6 months since completion of neo-adjuvant/adjuvant systemic therapy. The adjuvant/neoadjuvant therapy will be considered as 1 line of therapy
* Availability of tumor specimen for determination of PD-L1 and additional biomarker studies. Patient should be willing to undergo a pre-treatment biopsy as well as a biopsy after cycle 2 to evaluate the tumor microenvironment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients who have received prior treatment with anti-PD-1 or anti-PD-L1 inhibitors are eligible for the study
* Absolute neutrophil count >= 1,000/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 2 x upper limit of normal (ULN) or =< 3 x ULN for subjects with Gilbert's disease or liver metastases
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (=< 5 x ULN if evidence of hepatic involvement by malignant disease)
* Estimated glomerular filtration rate (eGFR) >= 40 mL/min/1.73m^2
* Lactate dehydrogenase (LDH) < 2 x ULN
* Provision of signed and dated informed consent form
* Life expectancy >= 3 months, as determined by the investigator
* Patients must have clinically and/or radiographically documented measurable disease. At least one site of disease must be uni-dimensionally measurable as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen during the 14 days prior to initiation of study treatment
* Subjects with central nervous system (CNS) metastases treated with radiation therapy (whole-brain radiation therapy [WBXRT] or stereotactic radiosurgery [SRS]) are eligible if, > 28 days following completion of radiation therapy (XRT), they show stable disease on post-treatment magnetic resonance imaging (MRI)/computed tomography (CT), are off corticosteroids, and are neurologically stable
* Female patients of childbearing potential have a negative pregnancy test at baseline. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti estrogens, or ovarian suppression

  * Patients who are not postmenopausal (>= 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within 14 days of treatment initiation
  * Sexually active women of childbearing potential enrolled in the study must agree to use 2 forms of accepted methods of contraception during the course of the study and for 12 weeks after their last dose of study drug. Effective birth control includes (a) intrauterine device plus 1 barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner

Exclusion Criteria:

* Subjects who have received 4 or more lines prior treatment in the metastatic setting
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Vitiligo, alopecia, hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, celiac disease controlled by diet alone or conditions not expected to recur in the absence of an external trigger are permitted
* History of psychiatric illness or social situations that would limit compliance with study requirements. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known active, untreated central nervous system (CNS) metastases and/or carcinomatous meningitis except for patients with =< 3 small (< 0.6 cm) asymptomatic brain lesions where treatment is not indicated. Patients with neurological symptoms must undergo a head computed tomography (CT) scan or brain magnetic resonance imaging (MRI) to exclude brain metastasis
* Subjects previously treated with pelareorep
* Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis
* Prior allogeneic stem cell or solid organ transplantation
* Patients may not have non-oncology vaccine therapies for prevention of infectious disease (for example, seasonal live influenza vaccine, human papilloma virus vaccine) within 4 weeks of study drug administration. Vaccination while on study is also prohibited except for administration of the inactivated influenza vaccine
* Known history of human immunodeficiency virus (HIV) or other serious immunocompromised state
* Known positive hepatitis B surface antigen undergoing anti-viral treatment and/or active hepatitis C indicated by positive quantitative hepatitis C virus (HCV) ribonucleic acid (RNA)
* Patient is pregnant or breastfeeding
* Receipt of any investigational treatment or anti-cancer therapy within 14 days of enrollment into the study
* Known hypersensitivity to the study drugs or their components
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) class III-IV within 6 months prior to their first dose of study drugs
* Prior malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 1 year prior to study entry
* Active alcohol or drug abuse per treating physician
* Patients may not participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial, throughout the duration of this study
* Toxicity of prior therapy that has not recovered to =< grade 1 or baseline (with the exception of any grade of alopecia and anemia not requiring transfusion support)
* For patients who have received prior immune-checkpoint therapy: Immune-related toxicity during prior checkpoint inhibitor therapy for which permanent discontinuation of therapy was recommended (per product label or consensus guidelines), OR any immune-related toxicity that required intensive or prolonged immunosuppression. (With the exception of endocrinopathy that is well controlled on replacement hormones)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Within 8 weeks after completion of treatment
  Defined as the percentage of participants having an objective response (complete response [CR] or partial response [PR]), according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The ORR of the drug will be assessed according to Simon's two stage design. The estimated ORR will be compared to the response rate specified in the null hypothesis (6%) using one-sided exact binomial test at type I error 5%. 95% confidence interval (C.I.) will be also reported.
Incidence of adverse events | Up to 2 years after completion of treatment
  Will be determined by the number, frequency, duration, and severity of adverse events (AEs) using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0; laboratory tests and vital signs.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the start of therapy until disease progression, or death due to any cause, assessed up to 2 years after completion of treatment
  Will be determined by the immune complete response (iCR). Will be estimated using Kaplan-Meier product-limit method. The median PFS times with two-sided 95% CIs will be estimated.
Overall survival (OS) | From the start of therapy until death due to any cause, assessed up to 2 years after completion of treatment
  Will be estimated using Kaplan-Meier product-limit method. The median OS times with two-sided 95% CIs will be estimated.
Duration of Response (DOR) | Up to 2 years after completion of treatment
  Defined as the time from an initial objective response (CR or PR) according to RECIST v 1.1 until disease progression, or death due to any cause, as determined by iCR.
Quality of life will be evaluated by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Core 30 (C30). | Up to 2 years after completion of treatment

OTHER OUTCOMES:
Changes in PD-L1 expression | Pre and post-treatment
  Will be correlated with treatment response.
T-cell receptor (TCR) sequencing | Up to 2 years after completion of treatment
  Assess the role of TCR sequencing in predicting treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Mridula A George, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Ohio State University Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes